CLINICAL TRIAL: NCT03871517
Title: INdobufen Versus aSpirin in acUte Ischemic stRokE,INSURE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Yongjun Wang, Executive Vice-President, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KY 2018-075-02
Record Dates: First submitted 2019-03-04; First posted 2019-03-12 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: Ischemic Stroke; Indobufen; Aspirin
MeSH Terms: conditions — Ischemic Stroke | interventions — indobufen; Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Indobufen (Experimental): Drug: Indobufen and aspirin mimetic Day 1 to 90±7: The first time : Indobufen 100mg + aspirin mimetic The second time: indobufen 100mg
  Interventions: Drug: Indobufen
- Aspirin (Active Comparator): Drug: Aspirin and Indobufen mimetic Day 1 to 90±7: The first time : aspirin 100mg+ Indobufen mimetic, The second time: indobufen mimetic.
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Indobufen — Indobufen inhibits platelet aggregation by reversibly inhibiting the platelet cyclooxygenase enzyme thereby suppressing thromboxane synthesis.
  Arms: Indobufen
Drug: Aspirin — Aspirin is a salicylate (sa-LIS-il-ate). It works by reducing substances in the body that cause pain, fever, and inflammation.
  Arms: Aspirin

SUMMARY:
China has the largest burden of cerebrovascular disease in the world. About 60% to 80% of which are ischemic stroke. In recent years, stroke has replaced heart disease and tumor diseases as the first cause of death and disability in adult population. The primary purpose of this study is to evaluate the efficacy of indobufen treatment in reducing the risk of a 3-month new stroke (any type of stroke, including ischemic stroke and hemorrhagic stroke) for patients with moderate/severe ischemic stroke is not inferior to aspirin therapy.

DETAILED DESCRIPTION:
China has the largest burden of cerebrovascular disease in the world. About 60% to 80% of which are ischemic stroke. In recent years, stroke has replaced heart disease and tumor diseases as the first cause of death and disability in adult population. The primary purpose of this study is to evaluate the efficacy of indobufen treatment in reducing the risk of a 3-month new stroke (any type of stroke, including ischemic stroke and hemorrhagic stroke) for patients with moderate/severe ischemic stroke is not inferior to aspirin therapy. The study is a multicenter, randomized, double-blind, positive drug parallel control and non-inferiority clinical design.

Non-inferiority analysis was performed on the primary efficacy analysis, and both intent analysis (ITT) and compliance program set (PPS) were used for analysis. If the indobufen group was confirmed to be non-inferior to aspirin (control group), a superiority analysis was further performed to analyze whether the indobufen was superior to aspirin. At the same time, Kaplan-Meier curves were used to simulate the cumulative risk of stroke (ischemic or hemorrhagic) at 90-day follow-up, and the Cox proportional hazards model was used to calculate the hazard ratio (HR) and 95% confidence interval, Log-rank test was used to evaluate the treatment effect. All statistics will be two-sided with p<0.05 considered significant.

All patients who received study drugs and with at least one safety follow-up record will be included in the safety population. The data for safety evaluation included adverse reactions observed during the trial and changes in laboratory data before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Female or male aged≥18 years and<80years.
* Acute moderate/severe ischemic stroke, 4≤NIHSS（National Institute of Health stroke scale）≤18 at the time of randomization.
* Patients can be randomized within 72 hours of symptoms onset.
* Provision of informed consent prior to any study specific procedures. * Symptom onset is defined by the "last seen normal" principle

Exclusion Criteria:

* Diagnosis of intracerebral hemorrhage such as cerebral hemorrhage, subarachnoid hemorrhage, etc.
* Diagnosis of hemorrhage or other pathology, such as vascular malformation, tumor, abscess or other major non-ischemic brain disease (e.g., multiple sclerosis) on baseline head CT or MRI.
* Moderate to severe ischemic stroke induced by angioplasty/vascular surgery.
* Modified Rankin Scale Score>2 at randomization (pre-morbid historical assessment).
* History of aneurysm (including intracranial aneurysm or peripheral aneurysms).
* Clear indication for anticoagulation (presumed cardiac source of embolus, e.g., atrial fibrillation, atrial myxoma, prosthetic cardiac valves known or suspected endocarditis).
* History of Hemostatic disorder, systemic bleeding, thrombocytopenia or neutropenia.
* History of previous symptomatic non-traumatic intracerebral bleed or cerebral artery amyloidosis.
* Gastrointestinal (GI) bleed within the past 6 months before randomization.
* Major surgery within the past 3 months before randomization.
* Severe renal or hepatic insufficiency. (Severe hepatic insufficiency is defined as alanine aminotransferase (ALT) value>3 times normal upper limit or Aspartate aminotransferase (AST)>2 times normal upper limit; Severe renal insufficiency is defined as creatinine>2 times normal upper limit).
* Diagnosis or of acute coronary syndrome.
* Other antithrombotic therapy are required during the study, including antiplatelet therapy(such as open-labeled aspirin, GPIIb/IIIa inhibitors, clopidogrel, ticagrelor, prasugrel, dipyridamole, ozagrel, cilostazol, etc.) and anticoagulant therapy(such as warfarin, thrombin and factor Xa inhibitors, bivalirudin, hirudin, argatroban, heparin and low molecular heparin, etc.).
* Within randomized 24 hours prior to any venous or arterial thrombolysis, mechanical bolt, snake venom, defibrase, lumbrokinase, etc.
* Heparin or oral anticoagulants were used within 10 days of randomization.
* Have a history of drug or food allergy and are known to be allergic to the study drug ingredients
* Planned or likely revascularization (any angioplasty or vascular surgery) within the next 3 months (if clinically indicated, vascular imaging should be performed prior to randomization whenever possible)
* Anticipated requirement for long-term (>7 days) non-steroidal antiinflammatory drugs (NSAIDs).
* The blood pressure needs to be controlled within the range of 90mmHg/60mmHg to 220mmHg/120mmHg.
* Suffering from serious cardiopulmonary disease, the researchers believe that it is not suitable for this study
* Patients with life expectancy<3 months or patients who are unable to complete the study for other reasons.
* Women of childbearing age who are negative in pregnancy test but refuse to practice reliable contraception. Women who are pregnant or lactating.
* Involving in other investigational drug or device tests within the past 30 days before randomization.
* Inability of the patient to understand and/or comply with study procedures and/or follow-up due to mental illness, cognitive or emotional disorders

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5438 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Any new stroke event (ischemic stroke or hemorrhagic stroke) | 3 months after randomization
  To evaluate the efficacy of indobufen treatment in reducing the risk of a 3-month new stroke (any type of stroke, including ischemic stroke and hemorrhagic stroke) for patients with moderate/severe ischemic stroke is not inferior to aspirin therapy.
Severe or moderate bleeding | 3 months after randomization
  GUSTO definition

SECONDARY OUTCOMES:
Any new stroke event | 1 year after randomization
  ischemic stroke or hemorrhagic stroke
New vascular events | 1 year after randomization
  ischemic stroke, hemorrhagic stroke, myocardial infarction, or vascular death
New ischemic stroke events | within 3 months and 1 year after randomization
  New ischemic stroke events
modified Rankin Scale (mRS) score was compared between 0-2 and 3-6 in the two groups. | During the 3-month and 1-year follow-up
  The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. It has become the most widely used clinical outcome measure for stroke clinical trials. The scale runs from 0-6, running from perfect health without symptoms to death: 0 - No symptoms.1 - No significant disability. Able to carry out all usual activities, despite some symptoms.2 - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.3 - Moderate disability. Requires some help, but able to walk unassisted.4 - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.5 - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.6 - Dead. The mRS scores between 3 to 6 points are considered to be poor functional outcome.
The proportion of mRS scores between 3 to 6 points | 3 months and 1 year
  The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. It has become the most widely used clinical outcome measure for stroke clinical trials. The scale runs from 0-6, running from perfect health without symptoms to death: 0 - No symptoms.1 - No significant disability. Able to carry out all usual activities, despite some symptoms.2 - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.3 - Moderate disability. Requires some help, but able to walk unassisted.4 - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.5 - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.6 - Dead. The mRS scores between 3 to 6 points are considered to be poor functional outcome.
Changes in neurological impairment | 3 months after randomization
  changes in National Institutes of Health Stroke Scale (NIHSS) score at 3 months compared to baseline. The NIHSS is a tool used by healthcare providers to objectively quantify the impairment caused by a stroke. The NIHSS is composed of 11 items, each of which scores a specific ability between a 0 and 4. For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment. The individual scores from each item are summed in order to calculate a patient's total NIHSS score. The maximum possible score is 42, with the minimum score being a 0. Stroke severity: 0 No stroke symptoms;1-4 Minor stroke;5-15 Moderate stroke;16-20 Moderate to severe stroke;21-42 Severe stroke
Quality of life at 3 months and 1 year follow-up | 3 months and 1 year after randomization
  We will use the EQ-5D-5L scale to evaluate the quality of life. EQ-5D-5L is a standardized instrument for measuring generic health status. It has been widely used in population health surveys, clinical studies, economic evaluation and in routine outcome measurement in the delivery of operational healthcare. The EQ-5D-5L has five domain scales (mobility, self-care, usual activities, pain and discomfort, and anxiety and depression) and five levels for each domain.
The proportion of early lower extremity venous thrombosis. | 3 months after randomization
  The proportion of early lower extremity venous thrombosis.
All bleeding events | 3 months after randomization
  all bleeding: including severe or moderate hemorrhage, intracranial hemorrhage
death | 3 months after randomization
  death
Adverse events or serious adverse events | 3 months after randomization
  such as gastrointestinal reaction, gastrointestinal bleeding and renal impairment

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tian Tan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pan Y, Meng X, Yuan B, Johnston SC, Li H, Bath PM, Dong Q, Xu A, Jing J, Lin J, Jiang Y, Xie X, Jin A, Suo Y, Yang H, Feng Y, Zhou Y, Liu Q, Li X, Liu B, Zhu H, Zhao J, Huang X, Li H, Xiong Y, Li Z, Wang Y, Zhao X, Liu L, Wang Y; INSURE Investigators. Indobufen versus aspirin in patients with acute ischaemic stroke in China (INSURE): a randomised, double-blind, double-dummy, active control, non-inferiority trial. Lancet Neurol. 2023 Jun;22(6):485-493. doi: 10.1016/S1474-4422(23)00113-8. Epub 2023 Apr 27. PMID 37121237
- [Derived] Pan Y, Meng X, Chen W, Jing J, Lin J, Jiang Y, Johnston SC, Bath PM, Dong Q, Xu AD, Li H, Wang Y. Indobufen versus aspirin in acute ischaemic stroke (INSURE): rationale and design of a multicentre randomised trial. Stroke Vasc Neurol. 2022 Oct;7(5):457-461. doi: 10.1136/svn-2021-001480. Epub 2022 Apr 7. PMID 35393360